CLINICAL TRIAL: NCT03639376
Title: Salivary LL-37 and Periodontal Health in Children Exposed to Passive Smoking
Brief Title: Passive Smoking and LL-37 in Children
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Meltem Karsiyaka Hendek, Assistant Professor, Kırıkkale University
Other Study IDs: 2016/140
Record Dates: First submitted 2018-08-16; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Innate Immunity; Periodontal Health
Keywords: Children; Cotinine; LL-37; Passive smoking; Periodontal health; Saliva

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Passive smoking-exposed children: This group consists of children whose family members have smoked at home since the birth of the child.
- Passive smoking-unexposed children: This group consists of children whose family members have not smoked at home since the birth of the child.

SUMMARY:
This study investigates the salivary LL-37 in passive smoking-exposed and unexposed children and the association between salivary LL-37 levels and periodontal clinical parameters in these children.Unstimulated salivary samples were collected from 180 children (90 passive smoking-exposed and 90 passive smoking-unexposed)

DETAILED DESCRIPTION:
Diverse mechanisms conduce to the detrimental periodontal effects of passive smoking, including alteration of both microbial and host response factors.

Antimicrobial peptides are considered to be an important intermediate step in initiating an initial immune response against the microbial side of the oral gingival epithelium and in the transition to acquired immunity.

LL-37 has a wide antimicrobial activity against both cariogenic and periopathogenic bacteria and its role in maintaining oral health has recently been stated

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy children

Exclusion Criteria:

* Any medications known to affect defense system and periodontium
* The presence of orthodontic / intraoral appliance

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children were selected from patients referred to Kirikkale University, Faculty of Dentistry, and Department of Pediatric Dentistry
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-11; Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Antimicrobial Peptide | In the first 18 months of study
  LL-37 (pg/mL)

SECONDARY OUTCOMES:
Passive smoking measurement | In the first 18 months of study
  Cotinine (ng/mL)